CLINICAL TRIAL: NCT06208813
Title: Assigned Creatine Ingestion With Usual Diet or Usual Diet Alone.
Brief Title: Creatine Supplementation in Concussion Recovery
Acronym: CSCR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Temp-4061
Record Dates: First submitted 2023-10-03; First posted 2024-01-17 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Concussion, Brain
MeSH Terms: conditions — Brain Concussion | interventions — Creatine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Participants will consume their normal daily diet.
- Creatine supplementation (Experimental): The intervention group will consume their usual diet plus 5 grams of creatine for the first four days following the initial meeting, and then 3 grams of creatine once per day thereafter until asymptomatic.
  Interventions: Dietary Supplement: Creatine

INTERVENTIONS:
Dietary Supplement: Creatine — Creatine supplementation
  Arms: Creatine supplementation

SUMMARY:
The proposed study aims to compare concussion recovery in those supplementing creatine and those not supplementing creatine. Specific aim 1: To compare number of days until asymptomatic between those taking creatine vs. those not taking creatine following a concussion. Hypothesis: The investigators hypothesize that individuals taking creatine will become asymptomatic sooner than those not taking creatine.Specific aim 2: To compare typical concussion assessment scores (i.e., symptom score, mental status, neurocognition, balance, motor coordination, and visual performance) between those taking creatine vs those not taking creatine following a concussion once asymptomatic.Hypothesis: The investigators hypothesize that individuals taking creatine will have better symptom scores, balance, mental status, and neurocognition assessment scores than those not taking creatine once asymptomatic.

The investigators will calculate descriptive statistics for all demographic, days to asymptomatic, and concussion assessments. For specific aim 1, The investigators will calculate a t-test to determine if days to asymptomatic differed in those taking creatine vs. those not taking creatine. For specific aim 2, the investigators will calculate t-tests with Bonferonni corrections to determine if concussion assessment scores (Sport Concussion Office Assessment Tool-6 assessments, CNS Vital Signs, visual assessment) differed in those taking creatine vs. those not taking creatine.

DETAILED DESCRIPTION:
Our proposed study aims to compare concussion recovery in those supplementing creatine and those not supplementing creatine. Specific aim 1: To compare number of days until asymptomatic between those taking creatine vs. those not taking creatine following a concussion. Hypothesis: The investigators hypothesize that individuals taking creatine will become asymptomatic sooner than those not taking creatine. Specific aim 2: To compare typical concussion assessment scores (i.e., symptom score, mental status, neurocognition, balance, motor coordination, and visual performance) between those taking creatine vs those not taking creatine following a concussion once asymptomatic. Hypothesis: The investigators hypothesize that individuals taking creatine will have better symptom scores, balance, mental status, and neurocognition assessment scores than those not taking creatine once asymptomatic.

Once the research team is contacted about a potential injury, the investigators will ensure the participant meets inclusion criteria prior to meeting and schedule a meeting if meet inclusion criteria to explain study details, obtain informed consent, administer a symptom checklist (Sport Concussion Office Assessment Tool-5, SCOAT-6) and demographic questionnaire, and provide creatine. The investigators will use the following components of the SCAOT-6: Removal from play and description, (Current Injury; p. 652), Symptom Evaluation (p. 654-655), Verbal Cognitive Tests (p. 655), Digits Backwards (p. 656), Months in Reverse (p. 656), Orthostatic Vital Signs (p.657), Balance (p. 658), Timed Tandem Gait (p. 658), Complex Tandem Gait (p. 659), Dual Task Gait (p.659), Modified Vestibular/Ocular-Motor Screen (p. 660), Anxiety Screen (p. 660), Depression Screen (p. 660), sleep screen (p. 661), Delayed Word Recall (p. 662) (requires approximately 1 hour). Participants will be randomly assigned to the intervention or control group (10 participants targeted for each group; participant identification numbers will be predetermined and allocated once enrolled). The intervention group will consume their usual diet plus 5 grams of creatine for the first four days following the initial meeting, and then 3 grams of creatine once per day thereafter until asymptomatic. The control group will be asked to consume their usual diet and no creatine. The investigators will then remain in contact with the participant to ensure compliance, and assess when the participant is asymptomatic. When the investigators contact the participant will vary depending on recovery process (e.g., if a participant has high symptom burden, they may allow a few days between contact; whereas if a participant is nearing asymptomatic, they contact the participant more frequently).

Once the participant becomes asymptomatic, the investigators will meet to administer a SCAOT-6, a computerized neurocognitive assessment (CNS Vital Signs), visual assessment (King-Devick) and note days from injury to asymptomatic. CNS Vital Signs requires approximately 20-25 minutes and assesses the domains of verbal and visual memory, psychomotor speed, reaction time, complex attention, cognitive flexibility, processing speed, executive function, simple attention, and motor speed. King-Devick is a visual assessment asking participants to read three test cards with numbers as fast as possible without committing errors. The investigators anticipate the assessment requiring approximately 1.5 hours.

The investigators will calculate descriptive statistics for all demographic, days to asymptomatic, and concussion assessments. For specific aim 1, the investigators will calculate a t-test to determine if days to asymptomatic differed in those taking creatine vs. those not taking creatine. For specific aim 2, the investigators will calculate t-tests with Bonferonni corrections to determine if concussion assessment scores (SCOAT-6 assessments, CNS Vital Signs, visual assessment) differed in those taking creatine vs. those not taking creatine.

ELIGIBILITY:
Inclusion Criteria:

* 18-35 years old with a diagnosed concussion within 72 hours post-injury

Exclusion Criteria:

* Learning disability, renal disease, mental behavior or migraine history, and current creatine use or have not taken creatine in the past 6 weeks

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Days to asymptomatic | From date of injury until the date in which symptoms are no longer experienced as measured by a symptom assessment, assessed up to 100 weeks
  Days to asymptomatic

SECONDARY OUTCOMES:
Symptom evaluation - Sport Concussion Office Assessment Tool 6 | From date of injury until the date in which symptoms are no longer experienced as measured by a symptom assessment, assessed up to 100 weeks
  22 item symptom list rated on a scale of 0-6 (0=none, 6=severe).
Standardized Assessment of Concussion - Sport Concussion Office Assessment Tool 6 | From date of injury until the date in which symptoms are no longer experienced as measured by a symptom assessment, assessed up to 100 weeks
  Mental status assessment scored out of 45.
Orthostatic Vital Signs - Sport Concussion Office Assessment Tool 6 | From date of injury until the date in which symptoms are no longer experienced as measured by a symptom assessment, assessed up to 100 weeks
  Blood pressure (mmHG) measured standing and supine; dichotomized as abnormal or normal considering both assessments for a single score.
Orthostatic Vital Signs - Sport Concussion Office Assessment Tool 6 | From date of injury until the date in which symptoms are no longer experienced as measured by a symptom assessment, assessed up to 100 weeks
  Heart rate (BPM) measured standing and supine; dichotomized as abnormal or normal considering both assessments for a single score.
Balance Error Scoring System - Sport Concussion Office Assessment Tool 6 | From date of injury until the date in which symptoms are no longer experienced as measured by a symptom assessment, assessed up to 100 weeks
  Six stances completed on firm and foam surface (double leg, tandem, single leg stances). Errors counted including lifting hands off hips, opening eyes, 30 degrees of hip abduction, putting foot down in single leg stance, and/or remaining out of position for great than 5 seconds.
Timed Tandem Gait - Sport Concussion Office Assessment Tool 6 | From date of injury until the date in which symptoms are no longer experienced as measured by a symptom assessment, assessed up to 100 weeks
  Walking 3-metre-long line on firm surface heel-to-toe. Three trials completed measured in seconds, and average of trials used as measurement.
Complex Tandem Gait - Sport Concussion Office Assessment Tool 6 | From date of injury until the date in which symptoms are no longer experienced as measured by a symptom assessment, assessed up to 100 weeks
  Participants instructed to "walk heel-to-toe quickly five steps forward, then continue forward with eyes closed for five steps." Points are counted for each step off the line, 1 point for truncal sway or holding onto an object for support. Completed again backwards. Total points are included for a single score (forward plus backward points).
Dual Task Gait Cognitive Accuracy Score - Sport Concussion Office Assessment Tool 6 | From date of injury until the date in which symptoms are no longer experienced as measured by a symptom assessment, assessed up to 100 weeks
  Patients are instructed "Now, while you are walking heel-to-toe, I will ask you to recite the following words in reverse order/count backwards out loud by 7's/ recite the months of the year in reverse order." We will measure the cognitive accuracy score (number correct/number attempted).
Dual Task Gait Average Time - Sport Concussion Office Assessment Tool 6 | From date of injury until the date in which symptoms are no longer experienced as measured by a symptom assessment, assessed up to 100 weeks
  Patients are instructed "Now, while you are walking heel-to-toe, I will ask you to recite the following words in reverse order/count backwards out loud by 7's/ recite the months of the year in reverse order." We will measure the average time (seconds).
Vestibular/Ocular-Motor Screening Smooth Pursuits | From date of injury until the date in which symptoms are no longer experienced as measured by a symptom assessment, assessed up to 100 weeks
  Test the ability to follow a slowly moving target. The patient and the examiner are seated. The examiner holds a fingertip at a distance of 3 ft. from the patient. The patient is instructed to maintain focus on the target as the examiner moves the target smoothly in the horizontal direction 1.5 ft. to the right and 1.5 ft. to the left of midline. One repetition is complete when the target moves back and forth to the starting position, and 2 repetitions are performed. The target should be moved at a rate requiring approximately 2 seconds to go fully from left to right and 2 seconds to go fully from right to left. The test is repeated with the examiner moving the target smoothly and slowly in the vertical direction 1.5 ft. above and 1.5 ft. below midline for 2 complete repetitions up and down. Again, the target should be moved at a rate requiring approximately 2 seconds to move the eyes fully upward and 2 seconds to move fully downward. Symptoms measured on a scale of 0-6.
Vestibular/Ocular-Motor Screening Saccades Horizontal | From date of injury until the date in which symptoms are no longer experienced as measured by a symptom assessment, assessed up to 100 weeks
  The examiner holds two single points (fingertips) horizontally at a distance of 3 ft. from the patient, and 1.5 ft. to the right and 1.5 ft. to the left of midline so that the patient must gaze 30 degrees to left and 30 degrees to the right. Instruct the patient to move their eyes as quickly as possible from point to point. One repetition is complete when the eyes move back and forth to the starting position, and 10 repetitions are performed. Record: Headache, Dizziness, Nausea & Fogginess ratings after the test. Symptoms measured on a scale of 0-6.
Vestibular/Ocular-Motor Screening Saccades Vertical | From date of injury until the date in which symptoms are no longer experienced as measured by a symptom assessment, assessed up to 100 weeks
  Repeat the test with 2 points held vertically at a distance of 3 ft. from the patient, and 1.5 feet above and 1.5 feet below midline so that the patient must gaze 30 degrees upward and 30 degrees downward. Instruct the patient to move their eyes as quickly as possible from point to point. One repetition is complete when the eyes move up and down to the starting position, and 10 repetitions are performed. Record: Headache, Dizziness, Nausea & Fogginess ratings after the test. Symptoms measured on a scale of 0-6.
Vestibular/Ocular-Motor Screening Convergence | From date of injury until the date in which symptoms are no longer experienced as measured by a symptom assessment, assessed up to 100 weeks
  Measure the ability to view a near target without double vision. The patient is seated and wearing corrective lenses (if needed). The examiner is seated front of the patient and observes their eye movement during this test. The patient focuses on a small target (approximately 14 point font size) at arm's length and slowly brings it toward the tip of their nose. The patient is instructed to stop moving the target when they see two distinct images or when the examiner observes an outward deviation of one eye. Blurring of the image is ignored. The distance in cm. between target and the tip of nose is measured and recorded. Abnormal: Near Point of convergence ≥ 6 cm from the tip of the nose.
Vestibular/Ocular-Motor Screening Vestibular-Ocular Reflex Horizontal | From date of injury until the date in which symptoms are no longer experienced as measured by a symptom assessment, assessed up to 100 weeks
  The patient is asked to rotate their head horizontally while maintaining focus on the target. The head is moved at an amplitude of 20 degrees to each side and a metronome is used to ensure the speed of rotation is maintained at 180 beats/minute (one beat in each direction). One repetition is complete when the head moves back and forth to the starting position, and 10 repetitions are performed. Record: Headache, Dizziness, Nausea and Fogginess ratings 10 sec after the test is completed. Symptoms measured on a scale of 0-6.
Vestibular/Ocular-Motor Screening Vestibular-Ocular Reflex Vertical | From date of injury until the date in which symptoms are no longer experienced as measured by a symptom assessment, assessed up to 100 weeks
  The test is repeated with the patient moving their head vertically. The head is moved in an amplitude of 20 degrees up and 20 degrees down and a metronome is used to ensure the speed of movement is maintained at 180 beats/minute (one beat in each direction). One repetition is complete when the head moves up and down to the starting position, and 10 repetitions are performed. Record: Headache, Dizziness, Nausea and Fogginess ratings after the test. Symptoms measured on a scale of 0-6.
Vestibular/Ocular-Motor Screening Visual Motion Sensitivity Test | From date of injury until the date in which symptoms are no longer experienced as measured by a symptom assessment, assessed up to 100 weeks
  Test visual motion sensitivity and the ability to inhibit vestibular-induced eye movements using vision. The patient stands with feet shoulder width apart, facing a busy area of the clinic. The examiner stands next to and slightly behind the patient, so that the patient is guarded but the movement can be performed freely. The patient holds arm outstretched and focuses on their thumb. Maintaining focus on their thumb, the patient rotates, together as a unit, their head, eyes and trunk at an amplitude of 80 degrees to the right and 80 degrees to the left. A metronome is used to ensure the speed of rotation is maintained at 50 beats/min (one beat in each direction). One repetition is complete when the trunk rotates back and forth to the starting position, and 5 repetitions are performed. Record: Headache, Dizziness, Nausea & Fogginess ratings after the test. Symptoms measured on a scale of 0-6.
Anxiety Screen - Sport Concussion Office Assessment Tool 6 | From date of injury until the date in which symptoms are no longer experienced as measured by a symptom assessment, assessed up to 100 weeks
  Participants are asked to rate seven items on a 0-3 point Likert-scale (0=Not at all, 3=Nearly every day). Scores are totaled and categorized into 0-4=minimal anxiety, 5-9=mild anxiety, 10-14=moderate anxiety, 15-21=severe anxiety.
Depression Screen - Sport Concussion Office Assessment Tool 6 | From date of injury until the date in which symptoms are no longer experienced as measured by a symptom assessment, assessed up to 100 weeks
  Participants are asked to rate two items with a variety of item responses. Scores are totaled with a cutpoint being 3 for depression.
Sleep Screen - Sport Concussion Office Assessment Tool 6 | From date of injury until the date in which symptoms are no longer experienced as measured by a symptom assessment, assessed up to 100 weeks
  Participants are asked to rate five items on a 0-3 point Likert-scale (0=Not at all, 3=Nearly every day). Item responses are total then categorized with 0-4=normal, 5-7 mild, 8-10 moderate, 11-17 severe clinical sleep disorder.
Verbal memory - CNS Vital Signs | Will be measured once at the asymptomatic timepoint; From date of injury until the date in which symptoms are no longer experienced as measured by a symptom assessment, no more than 100 weeks after injury
  Measures how well subject can recognize, remember, and retrieve words. Calculated using VBM (verbal memory) Correct Hits Immediate + VBM Correct Passes Immediate + VBM Correct Hits Delay + VBM Correct Passes Delay).
Visual memory - CNS Vital Signs | Will be measured once at the asymptomatic timepoint; From date of injury until the date in which symptoms are no longer experienced as measured by a symptom assessment, no more than 100 weeks after injury
  Measures how well subject can recognize, remember, and retrieve geometric figures. Calculated VIM (visual memory) Correct Hits Immediate + VIM Correct Passes Immediate + VIM Correct Hits Delay + VIM Correct Passes Delay).
Psychomotor speed - CNS Vital Signs | Will be measured once at the asymptomatic timepoint; From date of injury until the date in which symptoms are no longer experienced as measured by a symptom assessment, no more than 100 weeks after injury
  Measures how well a subject perceives, attends, responds to visual-perceptual information, and performs motor speed and fine motor coordination. Calculated finger tapping test (FTT) Right Taps Average + FTT Left Taps Average + Symbol Digit Coding Test Correct Responses.
Reaction time - CNS Vital Signs | Will be measured once at the asymptomatic timepoint; From date of injury until the date in which symptoms are no longer experienced as measured by a symptom assessment, no more than 100 weeks after injury
  Measures how quickly the subject can react, in milliseconds, to a simple and increasingly complex direction set. Calculated by Stroop Test Complex Reaction Time Correct + Stroop Reaction Time Correct) / 2.
Complex attention - CNS Vital Signs | Will be measured once at the asymptomatic timepoint; From date of injury until the date in which symptoms are no longer experienced as measured by a symptom assessment, no more than 100 weeks after injury
  Measures one's ability to track and respond to a variety of stimuli over lengthy periods of time and/or perform mental tasks requiring vigilance quickly and accurately. Calculated by Stroop Commission Errors + Shifting Attention Test Errors + Continuous Performance Test Commission Errors + Continuous Performance Test Omission Errors
Cognitive Flexibility- CNS Vital Signs | Will be measured once at the asymptomatic timepoint; From date of injury until the date in which symptoms are no longer experienced as measured by a symptom assessment, no more than 100 weeks after injury
  Measures how well subject is able to adapt to rapidly changing and increasingly complex set of directions and/or to manipulate the information.Calculated with Shifting Attention Test Correct Responses - Shifting Attention Test Errors - Stroop Commission Error
Processing speed - CNS Vital Signs | Will be measured once at the asymptomatic timepoint; From date of injury until the date in which symptoms are no longer experienced as measured by a symptom assessment, no more than 100 weeks after injury
  Measures how well a subject recognizes and processes information i.e., perceiving, attending/responding to incoming information, motor speed, fine motor coordination, and visual-perceptual ability. Calculated with Symbol Digit Coding Correct Responses - Symbol Digit Coding Errors
Executive function - CNS Vital Signs | Will be measured once at the asymptomatic timepoint; From date of injury until the date in which symptoms are no longer experienced as measured by a symptom assessment, no more than 100 weeks after injury
  Measures how well a subject recognizes rules, categories, and manages or navigates rapid decision making. Calculated with Shifting Attention Test Correct Responses - Shifting Attention Test Errors
Simple Attention - CNS Vital Signs | Will be measured once at the asymptomatic timepoint; From date of injury until the date in which symptoms are no longer experienced as measured by a symptom assessment, no more than 100 weeks after injury
  Measures one's ability to track and respond to a single defined stimulus over lengthy periods of time while performing vigilance and response inhibition quickly and accurately. Calculated with Continuous Performance (CPT) Correct Responses minus CPT Commission Errors.
Motor Speed - CNS Vital Signs | Will be measured once at the asymptomatic timepoint; From date of injury until the date in which symptoms are no longer experienced as measured by a symptom assessment, no more than 100 weeks after injury
  Measures one's ability to perform movements to produce and satisfy an intention towards a manual action and goal. Calculated with Finger Tapping Test Right Taps Average + Finger Tapping Test Left Taps Average.
King-Devick Visual Assessment | Will be measured once at the asymptomatic timepoint; From date of injury until the date in which symptoms are no longer experienced as measured by a symptom assessment, no more than 100 weeks after injury
  Visual assessment; The King-Devick Test is a two-minute rapid number naming assessment in which an individual quickly reads aloud single digit numbers and evaluates impairments of eye movements, attention and language function; fastest assessment of three cards measured in seconds

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Weber Rawlins, Principal Investigator — San Diego State University
Locations (1):
- San Diego State University, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roschel H, Gualano B, Ostojic SM, Rawson ES. Creatine Supplementation and Brain Health. Nutrients. 2021 Feb 10;13(2):586. doi: 10.3390/nu13020586. PMID 33578876
- [Result] Broglio SP, Cantu RC, Gioia GA, Guskiewicz KM, Kutcher J, Palm M, Valovich McLeod TC; National Athletic Trainer's Association. National Athletic Trainers' Association position statement: management of sport concussion. J Athl Train. 2014 Mar-Apr;49(2):245-65. doi: 10.4085/1062-6050-49.1.07. Epub 2014 Mar 7. PMID 24601910
- [Result] Giza CC, Hovda DA. The new neurometabolic cascade of concussion. Neurosurgery. 2014 Oct;75 Suppl 4(0 4):S24-33. doi: 10.1227/NEU.0000000000000505. PMID 25232881
- [Result] Harmon KG, Clugston JR, Dec K, Hainline B, Herring S, Kane SF, Kontos AP, Leddy JJ, McCrea M, Poddar SK, Putukian M, Wilson JC, Roberts WO. American Medical Society for Sports Medicine position statement on concussion in sport. Br J Sports Med. 2019 Feb;53(4):213-225. doi: 10.1136/bjsports-2018-100338. PMID 30705232